CLINICAL TRIAL: NCT00271076
Title: Carotid Artery Plaque Intravascular Ultrasound Evaluation
Brief Title: CAPITAL: Carotid Artery Plaque Intravascular Ultrasound Evaluation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arizona Heart Institute (Other)
Collaborators: Volcano Corporation (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AHI # 1119; Volcano Therapeutics
Record Dates: First submitted 2005-12-29; First posted 2005-12-30 (Estimated); Last update posted 2007-10-25 (Estimated); Status verified 2007-10

CONDITIONS: Carotid Artery Disease
Keywords: CAD; CEA; CAS; IVUS; symptomatic; asymptomatic; Cerebral Protection Device; TIA; Stroke; plaque morphology
MeSH Terms: conditions — Carotid Artery Diseases; Stroke

INTERVENTIONS:
Procedure: IVUS
Device: CAS
Procedure: CEA

SUMMARY:
To assess the safety and feasibility of Volcano Corp Eagle Eye Gold Catheter system to correlate the presence and characteristic of carotid artery atherosclerotic disease with anatomic and histologic analysis.

DETAILED DESCRIPTION:
A Phase , single center, prospective safety and feasibility study in patients diagnosed with carotid artery disease requiring intervention (carotid endarterectomy(CEA) or carotid artery stenting (CAS) with distal protection) as determined by the attending physician per standard treatment guidelines. At the time of the procedure, patients will undergo peri-operative assessment of their carotid artery disease with the study device.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Patient must be:

Symptomatic with lesions >/= to 50% stenosis, or Asymptomatic with lesions of >/= to 75% stenosis in at least one carotid artery, specific to the internal carotid artery, common carotid artery or bifurcated region; documented through acceptable ultrasound studies, completed within 30 days of recruitment.

* For patients with bilateral carotid disease- procedures need to be staged greater than 30 days apart. The lesion that has a greater degree of stenosis will be considered as the index procedure.
* Women of childbearing potential must have a negative pregnancy test within 7 days prior to treatment.
* The patient is able to give informed consent.

Exclusion Criteria:

* The patient is experiencing a new (acute) neurologic event or has experienced a stroke within the last 30 days prior to enrollment.
* The patient has intracranial tumors, arterial vascular malformations >5mm, aneurysms or severe intracranial stenosis distal to the target lesion.
* Presence of thrombus at the target site or loose 'floating' debris as determined by duplex analysis and/or angiography.
* Existing hemorrhagic disease or coagulation problems creating inability to obtain homeostasis at entry site.
* The patient has an allergy to, or is unable to tolerate, heparin, concomitant medications (clopidogrel or ticlid, aspirin) or to nitinol metal.
* The patient has a history of or known reaction to radiocontrast agent (radiopaque dye) and is unable to be premedicated.
* Coumadin treatment that has continued during the 48 hours prior to enrollment and an INR above hospital normals (i.e. in the event of atrial fibrillation or prosthetic valve replacement).
* Hemodynamic instability at the time of intervention.
* Severe chronic renal insufficiency (plasma/ serum creatinine> 2.5 mg/dL) at the time of intervention, except in patients on dialysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2006-01; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Primary endpoint: the completion of plaque morphology assessment & correlation of in-vitro histology with in-vivo histology using the Eagle Eye Gold Catheter.

SECONDARY OUTCOMES:
Secondary endpoint: safety and feasibility of the catheter system with respect to the possibility of assisting with the selection of a carotid stent, the relevance of pre-stent ballooning and ultimately the best treatment modality.

CONTACTS AND LOCATIONS:
Overall Officials: Edward B Diethrich, M.D., Principal Investigator — Arizona Heart Institute; Grayson H Wheatley, M.D., Study Director — Arizona Heart Institute
Locations (1):
- Arizona Heart Institute, Phoenix, Arizona, United States